CLINICAL TRIAL: NCT03885908
Title: Feasibility and Effectiveness of Automated Geriatric Co-Management Program on Improving the Perioperative Care of Older Patients With Solid Mass or Nodule Suspicious for Cancer
Brief Title: Automated Geriatric Co-Management Program in Older Patients With Solid Mass or Nodule Suspicious for Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-066
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Automated Geriatric Co-Management Program; Perioperative Care; Solid mass; Nodule; 19-066
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized controlled trial study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person geriatric co-management group (Active Comparator): "In-person" geriatric consults to be done via telemedicine due to the current pandemic and consideration for patient safety.
  Interventions: Other: in-person geriatric co-management
- Automated geriatric co-management program group (Experimental)
  Interventions: Other: automated geriatric co-management

INTERVENTIONS:
Other: in-person geriatric co-management — The geriatrics service sees these patients for at least 2 postoperative days, if deemed clinically necessary by the geriatrician. During the inpatient hospital course, the geriatrics service will ensure the execution of preoperative recommendations and will discuss with the surgical team, who will act as a primary team, any additional recommendation in order to improve postoperative care. "In-person" geriatric consults to be done via telemedicine due to the current pandemic and consideration for patient safety.
  Arms: In-person geriatric co-management group
Other: automated geriatric co-management — Following completion of the eRFA, the summary of impairments as well as the recommendations generated by the study team (hard-copy or email) will be provided in real-time to the surgery team for their attention.
  Arms: Automated geriatric co-management program group

SUMMARY:
The purpose of this study is to find out if it is possible to use the automated geriatric co-management program to manage the participants care before, during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Solid mass or nodule suspicious for cancer
* Aged 65 or older
* Being considered for surgical resection of the solid mass or nodule, with anticipated hospital length of stay of at least two days,
* Completed the eRFA per routine care

Exclusion Criteria:

* Unable to read or comprehend English
* Not having a completed electronic Rapid Fitness Assessment within 2 months of surgery**Note) To avoid excluding patients based this item, patients have to complete another eRFA within two months of surgery.
* Being discharged in one day or earlier from the hospital.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Shahrokni, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In-person Geriatric Co-management Group | Automated Geriatric Co-management Program Group
Started | 11 | 9
Completed | 8 | 7
Not Completed | 3 | 2
Not completed — Patient deemed to be ineligible due to language preference | 1 | 0
Not completed — Patient became ineligible becasue she underwent neoaedjuvant chemotherapy before surgery. | 1 | 0
Not completed — Patient did not undergo surgery within 2 months of consent. | 1 | 1
Not completed — Patient unable to complete appointment - withdrawn from study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-person Geriatric Co-management Group | Automated Geriatric Co-management Program Group | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Median (Full Range); unit: years] | 75 [65 to 88] | 76 [65 to 80] | 76 [65 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Automated Geriatric Co-management Program
Description: percentage of recommendations that were followed by the surgery team
Time Frame: 2 years
Population: N/A data were not collected
Arm/Group | In-person Geriatric Co-management Group | Automated Geriatric Co-management Program Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | In-person Geriatric Co-management Group | Automated Geriatric Co-management Program Group
All-Cause Mortality (participants affected / at risk) | 3/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03885908/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03885908/ICF_000.pdf